CLINICAL TRIAL: NCT01737437
Title: Effect of Lidocaine Sprayed on Direct Laryngoscopy and Trachea on Hemodynamics During Endotracheal Intubation
Brief Title: Effect of Lidocaine Sprayed on Hemodynamics During Endotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: php1
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Neurosurgical Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- group L (Experimental): 10% Lidocaine was applied to the laryngoscope blade and 0.9% normal saline was applied to the trachea.
  Interventions: Drug: group L
- group C (Placebo Comparator): 0.9% normal saline was applied to trachea and laryngoscope blade in Group C.
  Interventions: Drug: group C
- group V (Experimental): 0.9% normal saline was applied to the laryngoscope blade and 10% Lidocaine was applied on trachea.
  Interventions: Drug: group V
- group LV (Experimental): 10% Lidocaine was applied on laryngoscope blade and trachea.
  Interventions: Drug: group LV

INTERVENTIONS:
Drug: group C — 0.9% normal saline was applied to trachea and laryngoscope blade
  Arms: group C
Drug: group L — 10% Lidocaine was applied to the laryngoscope blade and 0.9% normal saline was applied to the trachea.
  Arms: group L
Drug: group V — 0.9% normal saline was applied to the laryngoscope blade and 10% Lidocaine was applied on trachea.
  Arms: group V
Drug: group LV — 10% Lidocaine was applied on laryngoscope blade and trachea.
  Arms: group LV

SUMMARY:
A previous study demonstrated topical lidocaine spray on the larynx and the trachea is effective in reducing hemodynamic response to laryngoscopy and endotracheal intubation. In clinical practice, blind oropharyngeal application of lidocaine without aiding direct laryngoscopy can not assured that sprayed lidocaine effectively reaches the larynx and trachea. Therefore, direct laryngoscopy should be necessary to reach topical lidocaine to correct sites. Unfortunately, direct laryngoscopy itself can affect hemodynamics during spraying lidocaine. In this study, we will investigate an effect of lidocaine sprayed on direct laryngoscopy and the tracheal mucosa on hemodynamic change throughout intubation.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-60 years,
* ASA groups I or II

Exclusion Criteria:

* ASA III or IV,
* hypertension,
* anticipated difficult airway, and
* severe coronary and cerebrovascular diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
mean blood pressure, heart rate | baseline, at laryngoscope insertion, 60s after laryngoscope insertion, during intubation, one, two, three min after endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea